CLINICAL TRIAL: NCT01510275
Title: Efficacy on Combined Use of Respiratory Devices RESPILIFT® and RESPIVOL® in Adult Cardio-thoracic Surgery Patients. Randomized-controlled Study
Brief Title: Combined Use of Respiratory Devices After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Pineta Hospital (Other)
Responsible Party: Principal Investigator, Prof. Clini Enrico, Prof., Villa Pineta Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-02-2010
Record Dates: First submitted 2012-01-10; First posted 2012-01-16 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Dyspnea; Well Being
Keywords: cardio-thoracic surgery; patients; pulmonary volume; respiratory muscle performance
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Combined use of RESPIVOL® and RESPILIFT® (with resistive load)
  Interventions: Device: Combined use of RESPIVOL® and RESPILIFT®
- Control (Sham Comparator): Combined use of RESPIVOL® and RESPILIFT® (without resistive load)
  Interventions: Device: Combined use of RESPIVOL® and RESPILIFT®

INTERVENTIONS:
Device: Combined use of RESPIVOL® and RESPILIFT® — Active devices (combined) for 14 consecutive session, bid, for 15 minutes.
  Arms: Intervention
Device: Combined use of RESPIVOL® and RESPILIFT® — Sham devices (combined) (without resistive load)for 14 consecutive session, bid, for 15 minutes.
  Arms: Control

SUMMARY:
In a rehabilitation setting, respiratory muscle training with re-expansion techniques in patients following cardio-thoracic surgery represents a consolidated intervention. New devices called RESPILIFT® and RESPIVOl® improve deep inspiration and pulmonary volume with an effect on respiratory muscle performance and perceived dispnoea. The aim of the investigators study is to test the clinical efficacy of RESPILIFT® and RESPIVOl® in patients with a recent history of cardio-thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* recent cardio-thoracic surgery (< 30 days of admission)
* compliance to pulmonary rehabilitation program

Exclusion Criteria:

* clinical instability
* concomitant severe co-morbidities
* inability to use respiratory devices

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle performance | Change from Baseline in MEP at 6 months
  Change of MEP (Maximum Expiratory Pressure)measure

SECONDARY OUTCOMES:
Respiratory muscle performance | Enrollment (T0), Day 8 (T8), at the end (T14) and after 6 months (T6m)
  Change of MIP (Maximum Inspiratory Pressure)measure
Pulmonary volumes | Enrollment (T0), Day 8 (T8), at the end (T14) and after 6 months (T6m)
  Change of Static and dynamic volumes (FEV1,FVC,VC,IC,RV)
Pulmonary gas exchange | Enrollment (T0), at the end (T14) and after 6 months (T6m)
  Change of arterial oxygen(PaO2) and use of oxygen (FiO2) in terms of PaO2/FiO2
Perceived dispnoea, well being and thoracic pain | At enrollment (T0), every day during the treatment (T2,T4, T6, T8, T10, T12), at the end (T14) and after 6 months (T6m)
  Change of perceived dispnoea, well being and thoracic pain measured through validated Visual Analogic Scale (VAS)
Perceived quality of life | Enrollment (T0), at the end (T14) and after 6 months (T6m)
  Change of perceived quality of life through Saint George Respiratory Questionnaire (SGRQ), italian version

CONTACTS AND LOCATIONS:
Overall Officials: Enrico E Clini, MD, Study Director — University of Modena - Ospedale Villa Pineta
Locations (1):
- Villa Pineta Hospital, Modena, Modena, Italy

REFERENCES:
- [Derived] Crisafulli E, Venturelli E, Siscaro G, Florini F, Papetti A, Lugli D, Cerulli M, Clini E. Respiratory muscle training in patients recovering recent open cardiothoracic surgery: a randomized-controlled trial. Biomed Res Int. 2013;2013:354276. doi: 10.1155/2013/354276. Epub 2013 Jul 30. PMID 23984352